CLINICAL TRIAL: NCT01244659
Title: An Open Randomized Non-inferiority Study to Compare Safety and Efficacy of Immunosuppressive Regiments Using Tacrolimus From EMS and Prograf® in Post Renal Transplanted Patients
Brief Title: A Randomized Study Assess the Safety and Efficacy of Tacrolimus vs Prograf® in Renal Transplantation Treatment
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACEMS0410
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Renal Transplant
Keywords: Tacrolimus; Immunosuppressive Agents; Kidney transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus from EMS (Experimental): Group 1: Tacrolimus from EMS + Myfortic® + Steroids
  Interventions: Drug: Tacrolimus from EMS
- Prograf (Active Comparator): Group 2: Prograf® + Myfortic® + Steroids
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Tacrolimus from EMS — Tacrolimus initial dose of 0.2 mg/kg/day Myfortic®: 720 to 1440 mg/day Steroids: methylprednisolone: first dose 500mg, 250 mg at first day and 125mg at second day, reducing to 30mg after third day post transplantation.
  Arms: Tacrolimus from EMS
Drug: Prograf — Prograf initial dose of 0.2 mg/kg/day Myfortic®: 720 to 1440 mg/day Steroids: methylprednisolone: first dose 500mg, 250 mg at first day and 125mg at second day, reducing to 30mg after third day post transplantation.
  Arms: Prograf

SUMMARY:
Comparison of safety and efficacy of immunosuppressive regiments using tacrolimus from EMS and Prograf® in post renal transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old
* Patient is receiving kidney from live or death donor
* Kidney donor younger than 65 years old
* PRA ≤ 30%
* Negative pregnancy test for women
* Patient agreement to practice birth control
* Patient has been fully informed and has given written informed consent

Exclusion Criteria:

* HLA identical
* Patient multi-organ transplant recipient
* Any pathology or past medical condition that can interfere with this protocol
* Allergy or intolerance of any study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | day 1 to day 180
  Incidence of biopsy confirmed acute rejection

SECONDARY OUTCOMES:
Safety | day 1 to day 180
  1. Patient and graft survival
  2. Renal function control by Estimated Glomerular Filtration Rate
  3. Safety, including incidence of post-transplant infection, malignances, diabetes mellitus, hepatotoxicity, blood pressure control and lipidic profile evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Pinho, MD, Study Director — EMS
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil